CLINICAL TRIAL: NCT01434030
Title: Development of a Behavioral Observer for Type 1 Diabetes Mellitus
Acronym: Phase1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14956; R01DK085623 (NIH)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Observer (Other): Focus group methodology was chosen to obtain qualitative and quantitative data on participants' desire to use glucose advisory systems to manage their diabetes, their concerns about and desired features and functions of these systems, and their perceived confidence with behavioral event recording. At the outset of each interview, the personalized glucose advisory system (PGASystem) was described to participants as a system composed of a continuous glucose monitor (CGM) device and insulin pump, into which they would input daily information about their insulin, food, and physical activity. The system would then use their data to create personalized algorithms and advice about various aspects of their diabetes management, such as suggestions regarding bolus and basal rate dosing. The interview consisted of open-ended, multiple choice, and dichotomous questions.
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — Focus group methodology was chosen to obtain qualitative and quantitative data on participants' desire to use glucose advisory systems to manage their diabetes, their concerns about and desired features and functions of these systems, and their perceived confidence with behavioral event recording. At the outset of each interview, the personalized glucose advisory system (PGASystem) was described to participants as a system composed of a continuous glucose monitor (CGM) device and insulin pump, into which they would input daily information about their insulin, food, and physical activity. The system would then use their data to create personalized algorithms and advice about various aspects of their diabetes management, such as suggestions regarding bolus and basal rate dosing. The interview consisted of open-ended, multiple choice, and dichotomous questions.

SUMMARY:
Development of a bio-behavioral stochastic model-predictive controller (SMPC) for use as an artificial pancreas in T1DM requires fundamental behavioral and physiology studies, as well as translational modeling and engineering development. In order to be successful, closed-loop control in Type 1 Diabetes Mellitus (T1DM) must adapt to individual physiologic characteristics and to the behavioral profile of each person. An essential part of this adaptation is biosystem (patient) observation. The investigators propose to lay the foundation for a closed-loop control system which will include algorithmic observers of patients' behavior and metabolic state.

DETAILED DESCRIPTION:
This intensive descriptive study will follow 60 adults with T1DM who are currently experienced with insulin pump use for a two-week training period plus a one month active study period during which the DexCom SEVEN® PLUS Continuous Glucose Monitor (CGM) will be used in tandem with the OmniPod® Insulin Management System. The OmniPod® has a built in FreeStyle glucometer that allows tagging of food and activity-related treatment behaviors with each self-monitoring blood glucose (SMBG) value. The OmniPod® personal digital assistant (PDA) also stores information about insulin delivery and meal size in relation to the carbohydrate content. Parallel recording of CGM and behavioral data, as well as psychometric instruments will produce a rich synchronized data set for each person that will ultimately lead to the development of a behavioral event generator for use in future open-loop and closed-loop control algorithms for intelligent insulin dosing.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus (as defined by the American Diabetes Association criteria or judgment of a physician) for at least two years prior to the enrollment in the study.
* Use of an insulin pump to treat their diabetes for at least six months.
* Actively using a bolus calculator function with the current insulin pump with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor.
* Age 21 - 65 years. The investigators will not be studying children since the DexCom Seven® Plus is not approved for use in children. Adults over age 65 are likely to have medical exclusions for the follow-up Phase 2 study, which involves induced hypoglycemia.
* Willingness to participate in the study for 6 weeks wearing a DexCom Seven® Plus CGM and OmniPod® insulin pump, performing self-monitoring blood glucose (SMBG) with the integral FreeStyle glucometer 4 times per day (before meals and bedtime) in addition to SMBG required to calibrate the CGM or to validate a low or high BG alarm (<70 mg/dl or >300 mg/dl), and recording behavioral events by tagging SMGB values throughout the study with meal and activity descriptors.
* Willingness to avoid consumption of acetaminophen-containing products for the duration of the study.
* Demonstration of proper mental status and cognition for completion of the study.

Exclusion Criteria:

* Pregnancy
* Psychiatric disorders that would interfere with study tasks (e.g. mental retardation, substance abuse)
* History of a systemic deep tissue infection with methicillin-resistant staph aureus or Candida albicans
* Known bleeding diathesis or dyscrasia
* Active enrollment in another clinical trial
* Medical requirement for acetaminophen-containing products during the study period for more than 1 week
* Medical condition that would make operating a CGM or insulin pump difficult (e.g. blindness, severe arthritis, extensive scar tissue at sites where devices are inserted).
* Need for magnetic resonance imaging (MRI)/magnetic resonance angiogram (MRA) during the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris P Kovatchev, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia - Center for Diabetes Technology, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Shepard JA, Gonder-Frederick L, Vajda K, Kovatchev B. Patient perspectives on personalized glucose advisory systems for type 1 diabetes management. Diabetes Technol Ther. 2012 Oct;14(10):858-61. doi: 10.1089/dia.2012.0122. Epub 2012 Aug 2. PMID 22856588

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Observer
Started | 57
Completed | 56
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Observer: Behavioral: This is a field study that will investigate behavioral events (e.g. meals, exercise) in T1DM and daily glucose patterns using an insulin pump, continuous glucose monitoring (CGM) data, and frequent SMBG tagged with behavioral markers (recent food and activity). From these data, a learning algorithm - behavioral observer - will be able to track over time key recurrent elements, such as wake-up time, meals, exercise, and daily patterns of risks for hypo- or hyperglycemia. In future controllers, behavioral observation such as this will be used to forecast upcoming routine events, enabling open-loop and closed-loop control algorithms to deal with the probabilistic patterns of patients' self-treatment behavior.
Arm/Group | Behavioral Observer
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 23
HbA1c [Mean (Standard Deviation); unit: percent glycated hemoglobin] | 7.7 (1.2)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Time since diagnosis of Type 1 Diabetes
  years | 24.1 (11.0)

OUTCOME MEASURES:

1. Primary Outcome: Desire to Receive Advice From Personal Glucose Advisory System (PGASystem)
Description: The categories below indicate types of information that could be received from a PGASystem and the percentage of participants who stated that they would like to receive this type of information from a PGASystem.
Time Frame: 2 hour focus group
Measure: Number; unit: percentage of participants
Arm/Group | Behavioral Observer
Number analyzed (Participants) | 56
percentage of participants
  Correction Boluses | 100
  Basal Rates | 92.9
  Meal Boluses/Inuslin to Carb Ratios | 94.6
  Hypoglycemia Risk | 85.7

2. Secondary Outcome: Willingness to Follow PGASystem Advice
Description: The categories below indicate types of information that could be received from a PGASystem and the percentage of participants who stated that they would follow this type of advice from a PGASystem.
Time Frame: 2 hour focus group
Measure: Number; unit: percentage of participants
Arm/Group | Behavioral Observer
Number analyzed (Participants) | 56
percentage of participants
  Correction Boluses | 53.6
  Meal Boluses | 60.4
  Basal Rates | 44.2

ADVERSE EVENTS:
Arm/Group | Behavioral Observer
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes